CLINICAL TRIAL: NCT00017797
Title: Evaluation of Metabolic Complications Associated With Antiretroviral Medications in HIV-1-Infected Pregnant Women
Brief Title: Problems Associated With the Use of Anti-HIV Drugs in HIV-Infected Pregnant Women
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: ACTG A5084; AACTG A5084
Record Dates: First submitted 2001-06-12; First posted 2001-08-31 (Estimated); Last update posted 2006-08-07 (Estimated); Status verified 2006-08

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy Complications, Infectious; HIV-1; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Glucose Intolerance
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Control

SUMMARY:
The purpose of this study is to find out if HIV-infected pregnant women who take protease inhibitors (PIs) are more likely to have blood sugar problems than those who do not take PIs.

HIV-infected people generally are treated with a combination of different types of anti-HIV drugs, 1 of which is usually a PI. The same holds true for pregnant women, but not much is known about the use of these drugs in pregnancy. Blood sugar and liver problems caused by anti-HIV drugs in nonpregnant patients are well known but their effects in pregnancy are not. Also, certain physical changes brought about by pregnancy may affect the way drugs are handled in the body. There remains a need for further study into the use of anti-HIV drugs during pregnancy and their effect on the safety of the mother and baby.

DETAILED DESCRIPTION:
The dramatic impact of potent combination antiretroviral therapies on the course of HIV disease has made the use of PIs routine in the care of HIV-1-infected individuals. Combination therapy likewise has become the standard of care in pregnant individuals, even though information on use of these drugs during human pregnancy is limited. There are no published prospective evaluations of toxicities experienced by pregnant women on PI-containing antiretroviral regimens, despite findings of metabolic disturbances of glucose, fatty acids, and cholesterol, as well as lactic acidosis/hepatic steatosis in nonpregnant individuals treated with antiretrovirals. Gastrointestinal (GI) side effects also are well documented in nonpregnant individuals treated with PIs, but have not been systematically evaluated in pregnancy. In addition, the physiologic changes brought about by pregnancy may influence the pharmacokinetics, safety, and side effects of antiretroviral drugs. There remains a need for further evaluation of the use of antiretrovirals during pregnancy and their impact on maternal, fetal, and infant safety.

Patients are stratified according to whether or not they are on a PI-containing antiretroviral regimen and the number of weeks of gestation (26 weeks or less versus greater than 26 weeks). Patients are followed at 8-week intervals from the time of entry until delivery or pregnancy termination, with an additional visit at 12 weeks after delivery or pregnancy termination. All infants born to study participants are evaluated at the time of delivery (anthropometrics and HIV DNA PCR) and are seen again at the mothers' 12-week post-delivery visit. Glucose tolerance testing and other metabolic studies are performed serially during pregnancy and again postpartum. This is an observational study and drugs are not supplied. Patients receiving antiretroviral therapy must obtain their own medications.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are female and 13 years of age or older.
* Are between 20 and 34 weeks pregnant at study entry.
* Had an ultrasound performed at 16 or more weeks of pregnancy.
* Have consent of a parent or guardian if under 18 years of age. The father of the baby, if available, also must give consent.
* Have taken the same anti-HIV drugs, including a PI, during the 8 weeks just before study entry. If not taking a PI or any anti-HIV drug, must not have taken a PI during the 8 weeks just before study entry. Patients must carry on this way for the entire study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have diabetes. Patients who have had diabetes caused by pancreas problems or steroid use in the past, but now have normal blood sugar without having to take drugs or special diets, are allowed. Patients who have had blood sugar problems in a past pregnancy also are allowed.
* Had a serious infection or medical condition within 30 days before study entry.
* Are enrolled in another study which requires a lot of blood tests.
* Take, or have taken in the 6 weeks before study entry, any of the following drugs: hormones (growth hormone, testosterone, or steroids), thalidomide, interleukins or interferons, efavirenz, hydroxyurea, drugs to control blood sugar, and anti-cancer drugs.
* Take, or have taken in the year before study entry, steroids, e.g., prednisone, for more than 14 days in any 3-month period. Inhaled steroids and steroid creams/ointments are allowed.
* Take, or have taken in the 30 days before study entry, PIs with lovastatin or simvastatin (2 drugs that lower the amount of fat in the blood).
* Have an ultrasound showing a major abnormality in the baby.
* Have problems with their pregnancy and/or are expecting more than 1 baby.
* Abuse drugs or alcohol.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Livingston, Study Chair
Locations (40):
- United States (39):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - The Med Ctr Inc, Columbus, Georgia
  - Univ of Hawaii, Honolulu, Hawaii
  - Mt Sinai Hosp Med Ctr / Dept of Pediatrics, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Univ of Marlyand (Pediatric), Baltimore, Maryland
  - Brigham and Womens Hosp, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Hutzel Hospital, Detroit, Michigan
  - Children's Hosp of Michigan, Detroit, Michigan
  - Hennepin County Med Ctr, Minneapolis, Minnesota
  - Univ of Minnesota, Minneapolis, Minnesota
  - Washington Univ (St.Louis), St Louis, Missouri
  - St Peter's Med Ctr, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Jacobi Med Ctr, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Washington, Seattle, Washington
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- San Juan City Hosp, San Juan, Puerto Rico

REFERENCES:
- [Derived] Livingston EG, Cohn SE, Yang Y, Watts HD, Bardeguez AD, Jones TB, Smith LM, Umbleja T, McComsey GA. Lipids and lactate in human immunodeficiency virus-1 infected pregnancies with or without protease inhibitor-based therapy. Obstet Gynecol. 2007 Aug;110(2 Pt 1):391-7. doi: 10.1097/01.AOG.0000271210.79340.4c. PMID 17666616